CLINICAL TRIAL: NCT01838876
Title: A Phase 3, Long-term, Open-label Study of Safety and Tolerability of Cariprazine as Adjunctive Therapy in Major Depressive Disorder
Brief Title: Long-term Safety and Tolerability of Cariprazine as an Adjunctive Treatment to Antidepressant Therapy in Patients With Major Depressive Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Collaborators: Gedeon Richter Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RGH-MD-76
Record Dates: First submitted 2013-04-22; First posted 2013-04-24 (Estimated); Results first posted 2019-08-21 (Actual); Last update posted 2019-08-21 (Actual); Status verified 2019-07

CONDITIONS: Major Depressive Disorder
Keywords: Major Depressive Disorder; MDD; Depression
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — cariprazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Cariprazine + ADT (Experimental): Cariprazine, flexible dose (titrated to a dose of 3.0 milligrams (mg) adjusted to 1.5 mg or 4.5 mg based on investigator's judgment of response and tolerability), oral administration, once daily plus antidepressant drug therapy (ADT) for 26 weeks.
  Interventions: Drug: Cariprazine; Drug: Antidepressant Therapy (ADT)

INTERVENTIONS:
Drug: Cariprazine — Cariprazine capsules 0.5 mg, 1.0 mg, and 1.5 mg; Cariprazine doses 1.5, 3.0, or 4.5 mg/day (d); patients will be titrated to a starting dose of 3.0 mg/d. Patients can stay on 3.0 mg/d or the dose can be adjusted to 1.5 mg or 4.5 mg based on investigator's judgment of response and tolerability. Oral administration.
Drug: Antidepressant Therapy (ADT) — ADT such as citalopram, escitalopram, fluoxetine, sertraline, paroxetine, vilazodone, venlafaxine, desvenlafaxine, duloxetine or bupropion prescribed in accordance with its respective FDA approved package insert for each drug

SUMMARY:
The objective of this study is to evaluate the long-term safety and tolerability of cariprazine as an adjunctive treatment to antidepressant therapy (ADT) in patients with Major Depressive Disorder (MDD).

ELIGIBILITY:
Inclusion Criteria:

* Patients who have provided consent prior to any study specific procedures
* Meets the Diagnostic and Statistical Manual of Mental Disorders, 4th Edition, Text Revision (DSM-IV-TR) criteria for MDD
* New patients must have ongoing inadequate response to protocol allowed ADTs as reported in Antidepressant Treatment Response Questionnaire (ATRQ)
* For rollover patients from RGH-MD-72 [NCT01715805], completion of Study RGH-MD-72 (either double-blind or single-blind treatment periods) with continued ADT treatment.

Exclusion Criteria:

* Patients who do not meet the DSM-IV-TR criteria for MDD.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 442 (Actual)
Dates: Start 2013-04-29 (Actual); Primary Completion 2015-07-27 (Actual); Study Completion 2015-07-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Willie Earley, MD, Study Director — Allergan
Locations (90):
- United States (88):
  - Forest Investigative Site 032, Tucson, Arizona
  - Forest Investigative Site 109, Tucson, Arizona
  - Forest Investigative Site 105, Fayetteville, Arkansas
  - Forest Investigative Site 018, Little Rock, Arkansas
  - Forest Investigative Site 029, Little Rock, Arkansas
  - Forest Investigative Site 082, Garden Grove, California
  - Forest Investigative Site 107, Long Beach, California
  - Forest Investigative Site 104, National City, California
  - Forest Investigative Site 022, Newport Beach, California
  - Forest Investigative Site 004, Oceanside, California
  - Forest Investigative Site 078, Rancho Mirage, California
  - Forest Investigative Site 080, Redlands, California
  - Forest Investigative Site 113, San Diego, California
  - Forest Investigative Site 054, San Diego, California
  - Forest Investigative Site 007, San Diego, California
  - Forest Investigative Site 031, Temecula, California
  - Forest Investigative Site 048, Denver, Colorado
  - Forest Investigative Site 114, Norwich, Connecticut
  - Forest Investigative Site 037, Coral Springs, Florida
  - Forest Investigative Site 053, Fort Myers, Florida
  - Forest Investigative Site 023, Hallandale, Florida
  - Forest Investigative Site 071, Hialeah, Florida
  - Forest Investigative Site 006, Leesburg, Florida
  - Forest Investigative Site 112, Maitland, Florida
  - Forest Investigative Site 026, Miami, Florida
  - Forest Investigative Site 075, Miami, Florida
  - Forest Investigative Site 027, North Miami, Florida
  - Forest Investigative Site 074, North Miami, Florida
  - Forest Investigative Site 036, Oakland Park, Florida
  - Forest Investigative Site 051, Orlando, Florida
  - Forest Investigative Site 044, South Miami, Florida
  - Forest Investigative Site 008, Tampa, Florida
  - Forest Investigative Site 019, Winter Park, Florida
  - Forest Investigative Site 060, Atlanta, Georgia
  - Forest Investigative Site 024, Atlanta, Georgia
  - Forest Investigative Site 017, Marietta, Georgia
  - Forest Investigative Site 047, Smyrna, Georgia
  - Forest Investigative Site 070, Chicago, Illinois
  - Forest Investigative Site 013, Hoffman Estates, Illinois
  - Forest Investigative Site 063, Libertyville, Illinois
  - Forest Investigative Site 062, Maywood, Illinois
  - Forest Investigative Site 072, Naperville, Illinois
  - Forest Investigative Site 010, Oak Brook, Illinois
  - Forest Investigative Site 068, Skokie, Illinois
  - Forest Investigative Site 061, Indianapolis, Indiana
  - Forest Investigative Site 042, Lafayette, Indiana
  - Forest Investigative Site 065, Overland Park, Kansas
  - Forest Investigative Site 073, New Orleans, Louisiana
  - Forest Investigative Site 049, Gaithersburg, Maryland
  - Forest Investigative Site 077, Rockville, Maryland
  - Forest Investigative Site 110, Rockville, Maryland
  - Forest Investigative Site 046, Boston, Massachusetts
  - Forest Investigative Site 045, Natick, Massachusetts
  - Forest Investigative Site 103, Saint Charles, Missouri
  - Forest Investigative Site 106, Berlin, New Jersey
  - Forest Investigative Site 014, Toms River, New Jersey
  - Forest Investigative Site 058, Albuquerque, New Mexico
  - Forest Investigative Site 028, Brooklyn, New York
  - Forest Investigative Site 016, New York, New York
  - Forest Investigative Site 025, Staten Island, New York
  - Forest Investigative Site 076, The Bronx, New York
  - Forest Investigative Site 050, Durham, North Carolina
  - Forest Investigative Site 067, Bismarck, North Dakota
  - Forest Investigative Site 011, Cincinnati, Ohio
  - Forest Investigative Site 015, Cincinnati, Ohio
  - Forest Investigative Site 055, Columbus, Ohio
  - Forest Investigative Site 066, Mason, Ohio
  - Forest Investigative Site 064, Middleburg Heights, Ohio
  - Forest Investigative Site 038, Oklahoma City, Oklahoma
  - Forest Investigative Site 035, Oklahoma City, Oklahoma
  - Forest Investigative Site 039, Oklahoma City, Oklahoma
  - Forest Investigative Site 003, Portland, Oregon
  - Forest Investigative Site 052, Allentown, Pennsylvania
  - Forest Investigative Site 102, Norristown, Pennsylvania
  - Forest Investigative Site 059, Lincoln, Rhode Island
  - Forest Investigative Site 001, Charleston, South Carolina
  - Forest Investigative Site 079, Austin, Texas
  - Forest Investigative Site 005, Houston, Texas
  - Forest Investigative Site 108, The Woodlands, Texas
  - Forest Investigative Site 069, Wichita Falls, Texas
  - Forest Investigative Site 111, Murray, Utah
  - Forest Investigative Site 041, Charlottesville, Virginia
  - Forest Investigative Site 081, Bellevue, Washington
  - Forest Investigative Site 100, Bothell, Washington
  - Forest Investigative Site 043, Seattle, Washington
  - Forest Investigative Site 101, Middleton, Wisconsin
  - Forest Investigative Site 056, Milwaukee, Wisconsin
  - Forest Investigative Site 057, Waukesha, Wisconsin
- Puerto Rico (2):
  - Forest Investigative Site 033, San Juan
  - Forest Investigative Site 034, San Juan

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Rollover participants from Study RGH-MD-72 [NCT01715805] were eligible for this study if they had completed either the double-blind treatment or the continued-treatment periods. New patients were eligible if they had an ongoing inadequate response to a protocol-allowed antidepressant therapy (ADT).
Groups:
- Cariprazine + ADT: Cariprazine, flexible dose (titrated to a dose of 3.0milligrams (mg) adjusted to 1.5 mg or 4.5 mg based on investigator's judgment of response and tolerability), oral administration, once daily plus antidepressant drug therapy (ADT) for 26 weeks.
Period: Overall Study
Arm/Group | Cariprazine + ADT
Started | 442
Safety Population; Received Study Drug | 345
Entered Safety Follow-up Period | 287
Completed | 209
Not Completed | 233
Not completed — Adverse Event | 49
Not completed — Insufficient Therapeutic Response | 10
Not completed — Protocol Violation | 34
Not completed — Withdrawal of Consent | 33
Not completed — Lost to Follow-up | 21
Not completed — Study or Site Terminated by Sponsor | 1
Not completed — Reason not Specified | 7
Not completed — Did not meet eligibility criteria | 78

BASELINE CHARACTERISTICS:
Population: Safety Population included all participants in the enrolled population who took at least 1 dose of cariprazine in this study.
Groups:
- Cariprazine + ADT: Cariprazine, flexible dose (titrated to a dose of 3.0 mg adjusted to 1.5 mg or 4.5 mg based on investigator's judgment of response and tolerability), oral administration, once daily plus antidepressant drug therapy (ADT) for 26 weeks.
Arm/Group | Cariprazine + ADT
Number analyzed (Participants) | 345
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.7 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 249
  Male | 96
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 280
  Race: Black or African American | 54
  Race: Asian | 6
  Race: American Indian or Alaska Native | 1
  Race: Native Hawaiian or Other Pacific Islander | 1
  Race: Other | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 75
  Ethnicity: Non-Hispanic or Latino | 270

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) in the Treatment Period
Description: An adverse event (AE) is any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. An adverse event can therefore be any unfavorable and unintended sign (i.e. laboratory value), symptom, or disease temporally associated with the use of a medicinal product, whether or not related to the medicinal product. A TEAE is an AE that occurs or worsens after receiving study drug.
Time Frame: First dose of study drug to last dose of study drug in the 26-week Treatment Period and within 30 days of last dose of study drug for participants who did not participate in the 2-week Safety Follow-up Period (Up to 30 weeks)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Cariprazine + ADT
Number analyzed (Participants) | 345
Participants | 274

2. Primary Outcome: Number of Participants With Newly Emergent Adverse Events (NEAEs) in the Safety Follow-up Period
Description: An AE is any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. An adverse event can therefore be any unfavorable and unintended sign (i.e. laboratory value), symptom, or disease temporally associated with the use of a medicinal product, whether or not related to the medicinal product. A NEAE is a new AE that occurred during the 2-week Safety Follow-up Period.
Time Frame: 2 weeks following the 26-week Treatment Period
Population: Participants in the Safety Population, all participants in the enrolled population who took at least 1 dose of cariprazine in this study, who entered the Safety Follow-up period.
Measure: Count of Participants; unit: Participants
Arm/Group | Cariprazine + ADT
Number analyzed (Participants) | 287
Participants | 20

3. Primary Outcome: Number of Participants With Clinically Significant Changes From Baseline in Clinical Laboratory Parameters
Description: Clinical laboratory parameters included tests of hematology, chemistry, urinalysis and prolactin. The investigator assessed the results for clinical significance.
Time Frame: Baseline (Week 0) to up to 26 weeks in the Treatment Period
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Cariprazine + ADT
Number analyzed (Participants) | 345
Participants | 0

4. Primary Outcome: Number of Participants With Clinically Significant Changes From Baseline in Vital Sign Parameters
Description: Vital sign parameters included blood pressure, pulse rate, body mass index (BMI), weight, and waist circumference. The investigator assessed the results for clinical significance.
Time Frame: Baseline (Week 0) to up to 26 weeks in the Treatment Period plus a 2-week Safety Follow-up Period (Up to 28 weeks)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Cariprazine + ADT
Number analyzed (Participants) | 345
Participants | 0

5. Primary Outcome: Number of Participants With Clinically Significant Changes From Baseline in Electrocardiograms (ECG)
Description: A standard 12-lead ECG was performed. The investigator determined the clinical significance of the ECG findings using the central ECG interpretation laboratory report.
Time Frame: Baseline (Week 0) to up to 26 weeks
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Cariprazine + ADT
Number analyzed (Participants) | 345
Participants | 1

6. Primary Outcome: Number of Participants With Extrapyramidal Symptom (EPS)-Related TEAEs
Description: Extrapyramidal symptoms are drug-induced movement disorders such as dystonia, akathisia, parkinsonism, bradykinesia, tremor, and tardive dyskinesia.
Time Frame: First dose of study drug to last dose of study drug in the 26-week Treatment Period plus a 2-week Safety Follow-up Period or within 30 days of last dose of study drug for participants who did not participate in the Safety Follow-up Period (Up to 30 weeks)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Cariprazine + ADT
Number analyzed (Participants) | 345
Participants | 98

7. Primary Outcome: Number of Participants in the Most Severe Suicidal Ideation and Suicidal Behavior Recorded on the C-SSRS During the Treatment Period
Description: The Columbia-Suicide Severity Rating Scale (C-SSRS) is a clinician-rated instrument that reports the severity of both suicidal ideation and behavior. Suicidal ideation is classified on a 5-item scale: 1 (wish to be dead) to 5 (active suicidal ideation with specific plan and intent). The C-SSRS also captures information about the intensity of ideation, specifically the frequency, duration, controllability, deterrents, and reasons for the most severe types of ideation. Suicidal behavior is classified on a 5-item scale: 0 (no suicidal behavior to 4 (actual attempt). More than 1 classification can be selected provided they represent separate episodes.
Time Frame: Baseline (Lead-in study Baseline for roll-over participants and prior to first dose in this study for new participants) to Week 26 in this study
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Cariprazine + ADT
Number analyzed (Participants) | 345
participants
  No Suicidal Ideation | 308
  Suicidal Ideation | 37
  Suicidal Ideation with Specific Plan and Intent | 1
  Ideation,Some Intent to Act,without Specific Plan | 0
  Ideation,any Methods,without Intent to Act | 6
  Non-specific Active Suicidal Thoughts | 3
  Wish to be Dead | 27
  No Suicidal Behavior | 344
  Suicidal Behavior | 1
  Completed Suicide | 0
  Actual Suicide Attempt | 1

8. Primary Outcome: Number of Participants With Treatment-Emergent Ocular Events
Description: A TEAE is an AE that occurs or worsens after receiving study drug. Ocular events are adverse events related to the eye.
Time Frame: as for outcome 6
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Cariprazine + ADT
Number analyzed (Participants) | 345
Participants | 1

9. Primary Outcome: Change From Baseline in the Arizona Sexual Experiences Scale (ASEX) Score
Description: The ASEX is a participant-completed scale to evaluate overall sexual experiences over the previous 7 days consisting of 5 questions answered on a scale of 1 (best) to 6 (worst) for a total possible score of 3 to 30 (2 questions were only answered if the participant was sexually active in the past week), higher score indicates greater sexual dysfunction. There are different forms for males and females. A negative change from Baseline indicates improvement.
Time Frame: Baseline (Lead-in study Baseline for roll-over participants and prior to first dose of this study for new participants) to End of Treatment (Up to Week 26) in this study
Population: Participants from the Safety Population, all participants in the enrolled population who took at least 1 dose of cariprazine in this study, with data available for analysis at the given time-point.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Cariprazine + ADT (Female): Cariprazine, flexible dose (titrated to a dose of 3.0 mg adjusted to 1.5 mg or 4.5 mg based on investigators judgment of response and tolerability), oral administration, once daily plus antidepressant drug therapy (ADT) for 26 weeks for female participants.
- Cariprazine + ADT (Male): Cariprazine, flexible dose (titrated to a dose of 3.0 mg adjusted to 1.5 mg or 4.5 mg based on investigators judgment of response and tolerability), oral administration, once daily plus antidepressant drug therapy (ADT) for 26 weeks for male participants.
Arm/Group | Cariprazine + ADT (Female) | Cariprazine + ADT (Male)
Number analyzed (Participants) | 229 | 88
score on a scale
  Baseline | 20.1 (5.9) | 17.2 (5.5)
  Change from Baseline to the End of Treatment | -0.9 (4.4) | -0.1 (4.6)

ADVERSE EVENTS:
Time Frame: First dose of study drug to last dose of study drug in the 26-week Treatment Period plus a 2-week Safety Follow-up Period or within 30 days of last dose of study drug for participants who did not participate in the Safety Follow-up Period (Up to 30 weeks)
Arm/Group | Cariprazine + ADT
All-Cause Mortality (participants affected / at risk) | 2/345
Serious Adverse Events (participants affected / at risk) | 7/345
Other Adverse Events (participants affected / at risk) | 274/345
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cariprazine + ADT (N=345)
Blood creatine phosphokinase increased (Investigations) | 1
Completed suicide (Psychiatric disorders) | 1
Fall (Injury, poisoning and procedural complications) | 1
Pneumonia (Infections and infestations) | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1
Spinal cord injury (Injury, poisoning and procedural complications) | 1
Substance-induced psychotic disorder (Psychiatric disorders) | 1
Suicide attempt (Psychiatric disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cariprazine + ADT (N=345)
Nausea (Gastrointestinal disorders) | 21
Fatigue (General disorders) | 30
Nasopharyngitis (Infections and infestations) | 30
Weight increased (Investigations) | 34
Akathisia (Nervous system disorders) | 55
Headache (Nervous system disorders) | 40
Dizziness (Nervous system disorders) | 20
Sedation (Nervous system disorders) | 19
Anxiety (Psychiatric disorders) | 34
Insomnia (Psychiatric disorders) | 34
Restlessness (Psychiatric disorders) | 34

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.